CLINICAL TRIAL: NCT03745781
Title: Open-Label Placebo for Functional Dyspepsia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000294
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Intervention Model Description: Arm 1: open-label placebo Arm 2: treatment as usual control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- open-label placebo (Experimental): open-label placebo
  Interventions: Drug: Placebos
- treatment as usual (No Intervention)

INTERVENTIONS:
Drug: Placebos — placebo pills
  Arms: open-label placebo

SUMMARY:
The study is evaluating the efficacy of open-label placebo for the treatment of functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Functional Dyspepsia

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
dyspepsia severity on a VAS from 0-100 | 3 weeks
  How severe have your dyspepsia symptoms been over the past 7 days (on a VAS from 0-100)?

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No